CLINICAL TRIAL: NCT04873297
Title: Metoclopramide vs Placebo for Prevention of Pneumonia in Acute Stroke Patients Fed Via Nasogastric Tubes
Brief Title: Metoclopramide vs Placebo for Prevention of Pneumonia in Acute Stroke
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Responsible Party: Principal Investigator, Muhammad Hassan, Resident in Neurology, Shaheed Zulfiqar Ali Bhutto Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Metoclopramide in Stroke
Record Dates: First submitted 2021-04-29; First posted 2021-05-05 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Acute Stroke; Aspiration Pneumonia
MeSH Terms: conditions — Stroke; Pneumonia, Aspiration | interventions — Metoclopramide; Trimethoprim, Sulfamethoxazole Drug Combination; Water

STUDY DESIGN:
Intervention Model Description: After taking permission from the Hospital Ethical Committee this study will be conducted at the Neurology department of PIMS. After informed written consent, all patients admitted to the Neurology ward with acute stroke on the basis of the clinical and radiologic evidence as defined in the operational definition will undergo detailed history and neurological examination. Patients beings grouped into 2 subgroup via lottery method. One group is given metoclopramide and one group will be given placebo (normal saline). SPSS version 23 will be used for data analysis. Post stratification chi square test will be applied. P value ≤0.05 will be considered significant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metoclopramide Group (Experimental): One group will be given metoclopramide 10mg TDS
  Interventions: Drug: Metoclopramide 10mg
- Placebo Group (Placebo Comparator): This group will be given placebo (normal saline 10ml via NG TDS)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metoclopramide 10mg — Tab. Metoclopramide 10mg TDS via NG tube
  Other Names: Metomide; Metoclop
  Arms: Metoclopramide Group
Drug: Placebo — Placebo 10 ml of plain water Via NG
  Other Names: Water
  Arms: Placebo Group

SUMMARY:
Pneumonia is a major cause of mortality and morbidity in patients with acute stroke fed via nasogastric tubes and may be because of vomiting and gastro-esophageal regurgitation. The aim of the study was to assess whether regular treatment with metoclopramide, a D2-receptor antagonist with antiemetic and gastric prokinetic actions, could reduce the rate of pneumonia.

DETAILED DESCRIPTION:
Patients admitted with no signs of pneumonia within 7 days of stroke onset and 48 hours of insertion of a nasogastric tube will be recruited into a single-blind randomized placebo-controlled study who will admit in Neurology Department, PIMS. Participants will receive metoclopramide 10 mg or placebo 3 times daily via the nasogastric tube for 4 days. Clinical signs of pneumonia will be recorded on alternate days. Pneumonia will be diagnosed if the patient has relevant clinical signs, high inflammatory markers, and new infiltrates on the chest radiograph. A sample size of 106 patients is calculated, 53 patients in each group. Non-probability consecutive sampling will be used for recruitment of participants. Study duration will be six months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either gender.
2. Patients within 7 days of acute ischemic or hemorrhagic stroke confirmed by computed tomographic scan of the brain who required nasogastric feeds for >24 hours, and could be recruited within 48 hours of NGT insertion
3. Age above 13 years.

Exclusion Criteria:

* Patients with aspiration pneumonia at the time of presentation.
* Patients with a history of chronic neurodegenerative diseases that could affect swallowing (e.g. Parkinson disease and motor neuron disease)
* Poor postural control (unable to sit up for swallowing assessment).
* Esophageal disorders,
* Contraindications to metoclopramide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2021-05-02 (Actual); Primary Completion 2021-10-02 (Actual); Study Completion 2021-10-02 (Actual)

PRIMARY OUTCOMES:
Number of episodes of aspiration pneumonia | 7 days
  Number of episodes of aspiration pneumonia will be observed after treatment with metoclopramide.

SECONDARY OUTCOMES:
Number of participants with swallowing improved +NGT removed | 7 days
  During admission patient's swallowing with improved and NG tube removed.
Number of participants with treatment withdrawn and NGT removed | 7 days
  Patient's swallowing with improved and treatment withdrawn and NG tube removed.
New onset of Fever | 7 days
  Aspiraton pneumonia will be assess in terms of fever (>98.6F)
Leukocytosis | 7 days
  Aspiration pneumonia will be assess in terms of leukocytosis on blood counts [ TLC >12000/uL]
Aspiration Pneumonia | 7 days
  Treatment with metoclopramide in patients with acute stroke is hypothesized to prevent aspiration pneumonia and pneumonia will be assess in terms of new findings on chest x-ray of patients [The posterior segment of the upper lobes and the superior segment of the lower lobes are most commonly involved lung sites when aspiration occurs in a recumbent patient. In an erect patient, aspiration is more likely to involve bilateral basal segments, middle lobe, and lingula- new exudate, new pleural effusion and new infiltrates]

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Hassan, MD, Principal Investigator — Shaheed Zulfiqar Ali Bhutto Medical University
Locations (1):
- Shaheed Zulfiqar Ali Bhutto Medical University, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No